CLINICAL TRIAL: NCT06765902
Title: Open-Label, Phase 2 Clinical Trial of Pre-Surgery and Post-Surgery Immunotherapy With N-803, ETBX-071, and M-CENK in Combination With Surgery for Participants With High-Risk Prostate Cancer Pre-Prostatectomy.
Brief Title: Immunotherapy Before and After Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ResQ110A-PROS
Record Dates: First submitted 2024-12-23; First posted 2025-01-09 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2024-12

CONDITIONS: High-risk Prostate Cancer
Keywords: Prostate Cancer; High-risk prostate cancer; Immunotherapy; N-803; ETBX-071; M-CENK; Radical prostatectomy; Pre-surgery immunotherapy; Post-surgery immunotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ALT-803

STUDY DESIGN:
Intervention Model Description: The interventional model represents a sophisticated approach that leverages both established surgical techniques and cutting-edge immunotherapies, delivered in a carefully structured sequence, to address a challenging clinical problem. The inclusion of autologous cell therapy adds a level of personalization, while the standardized procedures and detailed assessments ensure robust and reliable data collection.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Standard of Care + Immunotherapy in addition to surgery. (Experimental): The experimental arm of this study is the treatment group receiving the combination of pre- and post-surgery immunotherapy with N-803, ETBX-071, and M-CENK in addition to surgery.
  Interventions: Drug: N-803; Drug: ETBX-071; Drug: M-CENK

INTERVENTIONS:
Drug: N-803 — A subcutaneous injection of an IL-15 superagonist.
Drug: ETBX-071 — A subcutaneous injection of a prostate-specific antigen (PSA) adenovirus vaccine.
Drug: M-CENK — An intravenous infusion of the patient's own NK cells that have been expanded and activated in a laboratory.

SUMMARY:
This Phase 2 clinical trial is testing a new immunotherapy combination (N-803, ETBX-071, M-CENK) for men with high-risk prostate cancer before and after prostate surgery. The goal is to see if this treatment improves cancer outcomes and is safe.

DETAILED DESCRIPTION:
This study is an open-label, Phase 2 clinical trial investigating the efficacy and safety of a three-part immunotherapy regimen in combination with surgery for men with high-risk prostate cancer who have not yet undergone a prostatectomy. The immunotherapy consists of three components:

N-803 (Nogapendekin Alfa Inbakicept): A soluble complex consisting of a modified human interleukin-15 (IL-15) variant bound to a human IL-15 receptor alpha subunit/human immunoglobulin G (IgG) Fc fusion protein. N-803 acts as a growth and activation factor for natural killer (NK) cells and effector and memory T-cells, enhancing their ability to kill cancer cells and stimulate an immune response. It is administered subcutaneously.

ETBX-071 (hAd5 [E1-, E2b-, E3-]-PSA Vaccine): A replication-defective human adenovirus serotype 5 vector modified to encode human prostate-specific antigen (PSA). This vaccine is designed to induce a cell-mediated immune response against PSA-expressing prostate cancer cells. It is administered subcutaneously.

M-CENK (Autologous Memory Cytokine-Enriched NK Cells): These are the patient's own NK cells that are collected through apheresis, expanded and activated ex vivo using cytokines (IL-12, IL-15, and IL-18) to enhance their cytotoxicity and IFN-γ production. The resulting M-CENK cells are then infused intravenously.

Study Design:

The study involves three main phases:

Pre-surgery Immunotherapy: Participants receive N-803, ETBX-071, and M-CENK according to a specific schedule for six weeks before undergoing prostatectomy.

Surgery: Participants undergo a radical prostatectomy.

Post-surgery Immunotherapy: Following surgery, participants receive four cycles of the same immunotherapy regimen (N-803, ETBX-071, and M-CENK) over a 24-week period. Some participants may also receive external beam radiation therapy (EBRT) post-surgery at the discretion of the investigator.

Endpoints:

The study will assess several endpoints, including:

Primary Endpoints: Event-free survival (EFS) and biochemical recurrence-free survival (bRFS) are the main measures of the treatment's effectiveness in preventing cancer recurrence.

Secondary Endpoints: These include the rate of PSA reduction within six months post-surgery and safety assessments (adverse events, serious adverse events, changes in vital signs and laboratory tests).

Exploratory Endpoints: These are additional measures to assess quality of life, sexual function, immune responses, and changes in the tumor microenvironment.

Patient Selection:

The study includes men with high-risk prostate cancer, defined by specific criteria related to PSA levels, Gleason score, and tumor stage. Participants must meet specific inclusion criteria and cannot have certain pre-existing conditions or prior treatments that might interfere with the study.

Follow-up:

Participants will be followed for up to five years after completing the treatment, with regular monitoring and assessments.

This detailed description provides a more comprehensive overview of the study's design, methodology, and objectives.

ELIGIBILITY:
Inclusion Criteria:

* Age: Must be 18 years or older.
* Consent: Able to understand and provide signed informed consent that complies with Institutional Review Board (IRB) or Independent Ethics Committee (IEC) guidelines.
* Diagnosis: Histologically confirmed prostate adenocarcinoma (unless a local pathologist's report shows consistent findings).
* Performance Status: Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life Expectancy: Must have a life expectancy of at least 10 years.
* Germline Testing: Must have undergone germline testing at the time of initial diagnosis (and at recurrence, if applicable).
* Metastasis: No evidence of soft tissue disease metastasis (visceral or lymph nodes) on CT/MRI scan.
* Autoimmune Disease: No active or organ-threatening autoimmune disease.
* High-Risk Prostate Cancer: Must have high-risk or very high-risk prostate cancer according to 2024 NCCN guidelines (PSA >20 ng/mL, or Gleason Grade Group ≥4, or ≥cT3a).
* Adequate Hematologic and Organ Function: Must meet specific criteria for absolute neutrophil count (ANC), lymphocyte count, platelet count, hemoglobin, INR or aPTT, AST, ALT, and alkaline phosphatase levels. Certain exceptions are made for participants with liver or bone metastases.
* Ability to Attend Visits: Must be able to attend required study visits and return for adequate follow-up.
* Contraception: If male and not surgically sterile, must agree to use effective contraception for up to 7 months after treatment.

Exclusion Criteria:

* Prior Prostate Treatments: Prior surgical, cryotherapy, or high-intensity focused ultrasound treatment for prostate cancer; prior orchiectomy or hormonal therapy (GnRH agonists, NSAA).
* Prior Anti-Androgen Therapy: Prior treatment with first-generation or second-generation androgen receptor (AR) inhibitors (e.g., bicalutamide, flutamide, nilutamide, cyproterone acetate; enzalutamide, apalutamide, or darolutamide).
* Organ Transplantation: Receipt of any organ transplantation (excluding those that don't require immunosuppression, like corneal or hair transplants).
* Corticosteroid Use: Chronic systemic corticosteroid administration (>14 days within 28 days before treatment initiation) except for topical, inhaled, or nasal corticosteroids.
* Active Autoimmune Disease: Active autoimmune disease (e.g., Addison's disease, Hashimoto's thyroiditis, systemic lupus erythematosus, Sjogren's syndrome, scleroderma, myasthenia gravis, Goodpasture syndrome, or active Graves' disease). Exceptions are made for those with a history of autoimmune disease that did not require systemic immunosuppression and does not threaten vital organ function.
* Medications Affecting Urinary Symptoms or PSA: Use of medications for urinary symptoms (5-alpha reductase inhibitors, alternative medications known to alter PSA levels) within 28 days prior to study initiation.
* Recent Major Surgery or Systemic Therapy: Major surgery or systemic therapy (including investigational therapies) within 28 days prior to study initiation.
* Allergic Reactions: History of allergic reactions to compounds with similar chemical or biological composition to the study drugs.
* Significant Cardiovascular or Cerebrovascular Disease: Clinically significant cardiovascular/cerebrovascular disease (e.g., stroke, myocardial infarction, unstable angina, congestive heart failure, serious cardiac arrhythmia, or uncontrolled hypertension) within six months prior to the first planned dose of study drugs.
* Intercurrent Medical Illness: Serious intercurrent medical illness that would interfere with participation.
* Infections: Active HIV, hepatitis B or C infection.
* Live Attenuated Vaccines: Administration of a live, attenuated vaccine within three weeks before study entry or anticipation that such a vaccine will be required during the study.
* Inability to Comply: The investigator deems the participant unable or unwilling to comply with study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2031-01-31 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | These are assessed from the date of surgery until the occurrence of disease recurrence (EFS) or biochemical recurrence (bRFS), or until the end of the five-year follow-up period.
  The length of time from surgery to the first occurrence of disease recurrence (biochemical failure, local/regional recurrence, distant metastasis) or death.
Biochemical recurrence-free survival (bRFS) | These are assessed from the date of surgery until the occurrence of disease recurrence (EFS) or biochemical recurrence (bRFS), or until the end of the five-year follow-up period.
  The length of time from surgery to the first evidence of biochemical recurrence (two sequential increases in PSA levels by >0.2 ng/ml within 3-4 weeks) or death.

SECONDARY OUTCOMES:
Rate of PSA reduction | Assessed within 6 months post-surgery.
  The percentage decrease in PSA levels within six months post-surgery.
Safety (AEs and SAEs) | Up to 260 weeks.
  Assessment of adverse events (AEs), serious adverse events (SAEs), and clinically important changes in laboratory values and vital signs.

OTHER OUTCOMES:
Quality of life (QoL): | Approximately 13 months
  Assessed using validated questionnaires (EPIC-26 and PROMIS).
Sexual function | Approximately 13 months
  Assessed using the Sexual Health Inventory for Men (SHIM)
Changes in immune subsets and antigen-specific immune responses | Approximately 13 months
  Measured at baseline and end of treatment.
Tumor microenvironment (TME) changes | Approximately 13 months
  The tumor microenvironment (TME) is the complex ecosystem of cells, molecules, and extracellular matrix that surrounds and interacts with tumor cells.
Circulating tumor DNA (ctDNA) | Approximately 13 months
  Levels measured to monitor minimal residual disease.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Brown, Study Chair — ImmunityBio, Inc.